CLINICAL TRIAL: NCT02365454
Title: Feasibility Clinical Study to Evaluate the Safety and Performance of the NEXUS™ Aortic Arch Stent Graft System
Brief Title: NEXUS™ Aortic Arch Stent Graft System First In Man Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP004.00
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Thoracic Aortic Arch Disease; Thoracic Aortic Aneurysm
Keywords: TAA
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thoracic Aortic Disease Single Arm Study (Experimental): Thoracic Aortic Disease treated by Stent Graft Placement
  Interventions: Device: Stent Graft Placement (Nexus)

INTERVENTIONS:
Device: Stent Graft Placement (Nexus) — The Nexus stent graft is introduced through a groin to the diseased location at the Aortic Arch. Depending on the patients anatomy and other medical considerations the physician may decide that blood flow to the sub-clavian artery and possibly also to the left carotid artery is required to be maintained via "surgical bypass grafting", either immediately, or a few days, before the implantation. In addition to the incision for introducing the investigational stent graft, two smaller access sites are required, one at the groin on the opposite side and on into the Right Arm to the Brachial Artery.
  This endovascular procedure will likely require full anesthesia. The entire procedure is assisted by an angiography imaging system.

SUMMARY:
A multicenter, prospective, open-label, non-randomized, interventional clinical study, sponsored by Endospan Ltd. Patients will be followed-up for five years.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and performance of the Nexus™ Aortic Arch Stent Graft System for the endovascular treatment of thoracic aortic pathologies requiring landing in the Aortic Arch (zone 0, zone 1, zone 2).

The Nexus™ Aortic Arch Stent Graft System is indicated for the endovascular treatment of thoracic aortic pathologies involving the aortic arch (such as aneurisms and dissections). The Nexus™ is intended to exclude the lesion from the blood circulation in patients diagnosed with thoracic aortic pathology and who have appropriate anatomy to accommodate the Nexus™ system in an endovascular procedure.

The primary objectives of the study are to evaluate the safety and performance of the Nexus™ Aortic Arch Aneurysm Stent Graft System.

ELIGIBILITY:
Inclusion Criteria:

* Male and female age ≥ 18.
* Any Thoracic Aorta pathology requiring landing in the Aortic Arch (zone 0, zone 1, zone2), e.g. aneurysm, dissection, false/Pseudo aneurysm.
* In patient with a thoracic aneurysm: dilatation of the aortic arch larger than 5.5cm in diameter, or symptomatic aneurysm of the aortic arch, or aortic diameter growth rate > 5mm per 6 months
* Patient is considered an appropriate candidate for an elective surgery, as evaluated by Physical Status Classification System I, II or III (American Society of Anesthesiologists).
* Femoral artery diameter as documented by CTA or MRA that allows endovascular access to the diseased site with a 20-22Fr delivery catheter.
* Access vessels morphology suitable for endovascular repair in terms of tortuosity, calcification and angulation, documented by CTA, MRA.
* Access vessel (femoral/iliac) diameter > 7 mm
* Ascending Aorta landing zone length > 30 mm
* Brachial/Axial Artery diameter > 3 mm
* Patient understands and is voluntarily willing to participate as evidenced by personally signing the Informed Consent document, and willingness to comply with follow-up schedule

Exclusion Criteria:

* Female is of childbearing potential
* Life expectancy of less than 1 year
* Any medical condition that, according to the investigator's decision, might expose the patient to increased risk by the investigational device or procedure.
* Acutely ruptured or instable aneurysm or an acute vascular injury due to trauma or infected penetrating ulcers of the aorta.
* Patient with an increased risk for aneurysm rupture during the procedure.
* Patient whose arterial access site is not anticipated to accommodate the access of the Nexus™ Delivery System, due to size, tortuosity or hostile groins (scarring, obesity, or previous failed puncture)
* Patients with severe atherosclerosis or intraluminal thrombus of the aorta or in the BCT
* Patient is suffering from unstable angina or NYHA classification III and IV and/or ASA classification IV and above.
* Patient has had a myocardial infarction (MI) or cerebral vascular accident (CVA) within 3 months prior to the planned implantation
* Patient has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment.
* Patient with a contraindication to undergo angiography
* Patient with known sensitivities or allergies to the device materials- Nitinol and polyester
* Clinical conditions that severely inhibit x-ray visualization of the Aorta.
* Connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndromes)
* Patient has history of bleeding diathesis or coagulopathy that may limit the use of dual antiplatelet or anticoagulant therapy by the decision of the investigator
* Patient has an active systemic infection at the time of the procedure documented by pain, fever, drainage, positive culture and/or leukocytosis (WBC > 11,000 mm3).
* Patients who have the condition that threatens to infect the stent graft.
* Acute renal failure; chronic renal failure (excluding dialysis); Creatinine > 2.00 mg/dl or > 182 umol/L
* Patient underwent major surgery or interventional procedure in the last three months.
* Any other medical, social, or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, or the procedures and evaluations pre- and post- treatment.
* Active participation in another clinical trial that is reasonable to conflict with the NexusTM study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Safety: Device related mortality at 30 days post implantation | 30 days

SECONDARY OUTCOMES:
Safety: Device related re-intervention within 1 year from implantation | 1 year

OTHER OUTCOMES:
Performance: Assess the rate of successful disease treatment at 30 days post implantation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lachat, Prof. MD, Principal Investigator — Klinic Hirslanden, Switzerland
Locations (4):
- Faculty Hospital Hradec Kralove, Hradec Králové, Czechia
- San Filippo Neri Hospital, Rome, Italy
- Switzerland (2):
  - Klinic Hirslanden, Zurich, Witellikerstrasse 40
  - Zurich University Hospital, Zurich